CLINICAL TRIAL: NCT05239338
Title: Preserving Fertility After Colorectal Cancer: The PREFACE Study
Brief Title: Preserving Fertility After Colorectal Cancer Study
Acronym: PREFACE
Status: Recruiting | Type: Observational
Sponsor: Andreana Holowatyj, PhD, MSCI (Other)
Responsible Party: Sponsor-Investigator, Andreana Holowatyj, PhD, MSCI, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Other Study IDs: VICC GI 2186
Record Dates: First submitted 2021-11-09; First posted 2022-02-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PREFACE: Vanderbilt-Ingram Cancer Center: Patient recruitment and follow-up, longitudinal collection of data and multiple biospecimen at pre-defined study timepoints, objective assessment of health behaviors/habits, individual interviews.

SUMMARY:
The PREFACE Study is a prospective, longitudinal cohort study of reproductive health and clinical outcomes among individuals diagnosed with colorectal cancer between age 18 to 49 years.

DETAILED DESCRIPTION:
The Preserving Fertility After Colorectal Cancer (PREFACE) Study comprehensively investigates fertility, sexual health and clinical outcomes along the cancer care continuum among individuals diagnosed with colorectal cancer between age 18 to 49 years.

Patients are recruited prior to colorectal cancer therapy [baseline] and followed for up to 36 months after completion of first-course therapy (or 45 months after diagnosis for patients on maintenance therapy). Study timepoints are defined at: (i) completion of first-course treatment (or 9 months after diagnosis for patients on maintenance therapy [treatment]); (ii) and at 9, 18 and 36 month intervals thereafter [surveillance]. This cohort is enriched by a robust collection of biospecimens and data.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of colorectal cancer
* Age 18 to 49 years at colorectal cancer diagnosis
* Diagnosed by and/or consulting with a physician participating in the PREFACE Study
* No prior history of colorectal cancer and/or colorectal cancer treatment
* Mentally and physically able to consent and participate in the study

Exclusion Criteria:

* Women who are pregnant at the time of colorectal cancer diagnosis
* Prisoners
* Unable to provide informed consent
* Unable to read, write, or complete questionnaires in English

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals diagnosed with colorectal cancer between the ages of 18 to 49 years.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2036-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Change(s) in serum hormonal markers | Baseline, treatment and multiple surveillance timepoints (up to 5 years)
  For female patients not taking oral contraceptive pills (OCPs), serum hormonal markers to be measured include: anti-Mullerian hormone (AMH), estrogens, sex hormone binding globulin (SHBG), follicle-stimulating hormone (FSH), luteinizing hormone (LH) and androgens. For male patients, serum hormonal markers to be measured include: inhibin B, FSH, androgens, estrogens, SHBG and LH.
Reproductive health history (Questionnaire) | Baseline timepoint
Change(s) in reproductive health (Questionnaire) | Baseline, treatment and multiple surveillance timepoints (up to 5 years)
Sexual health history (Questionnaire) | Baseline timepoint
Changes in sexual health (Questionnaire) | Baseline, treatment and multiple surveillance timepoints (Up to 5 years)
Sexual health (Interview) | 9 month post-treatment/Surveillance timepoint
Disease-free survival | Up to 5 years

SECONDARY OUTCOMES:
Change(s) in health-related quality of life (Questionnaire) | At baseline, treatment and multiple surveillance timepoints (Up to 5 years)
Physical activity (Accelerometer) | Baseline timepoint
Physical activity (Accelerometer) | Completion of first-course treatment (or 9 months after baseline)
Physical activity (Accelerometer) | 9 month post-treatment/Surveillance timepoint
Physical activity (Accelerometer) | 18 month post-treatment/Surveillance timepoint
Physical activity (Accelerometer) | 36 month post-treatment/Surveillance timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Andreana N Holowatyj, PhD, MSCI, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Holowatyj AN, Eng C, Lewis MA. Incorporating Reproductive Health in the Clinical Management of Early-Onset Colorectal Cancer. JCO Oncol Pract. 2022 Mar;18(3):169-172. doi: 10.1200/OP.21.00525. Epub 2021 Sep 23. No abstract available. PMID 34554830
- [Background] Eng C, Jacome AA, Agarwal R, Hayat MH, Byndloss MX, Holowatyj AN, Bailey C, Lieu CH. A comprehensive framework for early-onset colorectal cancer research. Lancet Oncol. 2022 Mar;23(3):e116-e128. doi: 10.1016/S1470-2045(21)00588-X. Epub 2022 Jan 31. PMID 35090673
- [Background] Keller SR, Rosen A, Lewis MA, Park HK, Babyak R, Feldman J, Ye F, Agarwal R, Ciombor KK, Geiger TM, Eng C, Hunzinger KJ, Viskochil RH, Roach MK, Velez Edwards DR, Cote ML, Holowatyj AN. Patient-Reported Discussions on Fertility Preservation Before Early-Onset Cancer Treatment. JAMA Netw Open. 2024 Nov 4;7(11):e2444540. doi: 10.1001/jamanetworkopen.2024.44540. PMID 39531236
- See also: PREFACE Study Website — http://www.theprefacestudy.org